CLINICAL TRIAL: NCT00607490
Title: Cognitive-behavioral Therapy for Vulvodynia: a Clinical Trial
Brief Title: A Randomized Clinical Trial for Women With Vulvodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Robin Masheb, Yale University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HD038493 (NIH)
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2008-01

CONDITIONS: Vulvodynia
Keywords: Vulvodynia; Vulvar pain; Dyspareunia; Sexual dysfunction; Vestibulitis
MeSH Terms: conditions — Vulvodynia; Dyspareunia; Sexual Dysfunction, Physiological | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-behavioral Therapy (Experimental): 10 weekly individual 60-minute sessions
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- Supportive Psychotherapy (Active Comparator): 10 weekly individual 60-minute sessions
  Interventions: Behavioral: Supportive Psychotherapy

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy — Behavioral, cognitive, sex therapy and relaxation interventions administered to teach self-management skills for pain control.
  Arms: Cognitive-behavioral Therapy
Behavioral: Supportive Psychotherapy — Patient-centered talk therapy to assist participants in expressing their thoughts and feelings.
  Arms: Supportive Psychotherapy

SUMMARY:
This study will evaluate the relative effectiveness of cognitive-behavioral therapy and supportive psychotherapy for the treatment of women with vulvodynia.

DETAILED DESCRIPTION:
Many treatments used for women with vulvodynia are based solely upon expert opinion. This randomized trial aimed to test the relative efficacy of cognitive-behavioral therapy (CBT) and supportive psychotherapy (SPT) in women with vulvodynia. Of the 50 participants, 42 (84%) completed 10-week treatments and 47 (94%) completed one-year follow-up. Mixed effects modeling was used to make use of all available data. Participants had statistically significant decreases in pain severity (p's<.001) with 42% of the overall sample achieving clinical improvement. CBT, relative to SPT, resulted in significantly greater improvement in pain severity during physician examination (p=.014), and greater improvement in sexual function (p=.034), from pre- to post-treatment. Treatment effects were well maintained at one-year follow-up in both groups. Participants in the CBT condition reported significantly greater treatment improvement, satisfaction and credibility than participants in the SPT condition (p's<.05). Findings from the present study suggest that psychosocial treatments for vulvodynia are effective. CBT, a directed treatment approach that involves learning and practice of specific pain-relevant coping and self-management skills, yielded better outcomes and greater patient satisfaction than a less directive approach.

ELIGIBILITY:
Inclusion Criteria:

* Independently diagnosed with vulvodynia by two study physicians

Exclusion Criteria:

* Any conditions known to better account for the vulvar pain
* Psychotic illness
* Actively suicidal
* Substance dependent
* Life-threatening illness
* Initiated psychotherapy, psychopharmacologic treatment or pain medication within one month prior to beginning the assessment phase of the study.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2000-09; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Pain Severity | Measured at 1-year follow-up

SECONDARY OUTCOMES:
Sexual Functioning | Measured at 1-year follow-up
Emotional Functioning | Measured at 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Robin M Masheb, Ph.D., Principal Investigator — Yale University